CLINICAL TRIAL: NCT02728583
Title: The Effects of a Low-fat Spread With Added Plant Sterol Esters and Fish Omega-3 Fatty Acids on Blood Lipids
Brief Title: The Effects of a Spread With Added Plant Sterols and Omega-3 Fatty Acids on Blood Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-SCC-2150
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Vascular Diseases; Hypercholesterolemia
Keywords: Plant sterols; Fish oil; Blood lipids
MeSH Terms: conditions — Vascular Diseases; Hypercholesterolemia | interventions — Phytosterols; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Margarine enriched with plant sterols and fish oil (Active Comparator): Low-fat margarine (25 g per day) with added plant sterols and Eicosapentaenoic acid (EPA) + Docosahexaenoic acid (DHA) from fish oil
  Interventions: Dietary Supplement: Margarine enriched with plant sterols and fish oil
- Placebo margarine (Placebo Comparator): Low-fat margarine (25 g per day) without added plant sterols and EPA + DHA
  Interventions: Dietary Supplement: Placebo margarine

INTERVENTIONS:
Dietary Supplement: Margarine enriched with plant sterols and fish oil
  Arms: Margarine enriched with plant sterols and fish oil
Dietary Supplement: Placebo margarine
  Arms: Placebo margarine

SUMMARY:
The main aim of the study is to investigate the effect of daily consumption of a margarine enriched with plant sterol esters and fish oil on fasting triglycerides (TG) concentrations.

The study also aims to investigate the effect of plant sterols and fish oil on fasting total cholesterol (TC), Low-density lipoprotein cholesterol (LDL-C), High-density lipoprotein cholesterol (HDL-C) and non-HDL-C.

At last, the effect of plant sterols and fish oil on fasting apolipoprotein concentrations will be explored.

DETAILED DESCRIPTION:
The main aim of the study is to investigate the effect of daily consumption of a margarine enriched with plant sterol esters and fish oil on fasting TG concentrations.

The study also aims to investigate the effect of plant sterols and fish oil on fasting TC, LDL-C, HDL-C and non-HDL-C.

At last, the effect of plant sterols and fish oil on fasting apolipoprotein concentrations will be explored. This exploratory objective will only be analyzed if a relevant treatment effect on fasting triglycerides concentrations is observed.

ELIGIBILITY:
Inclusion Criteria:

* Fasting TG levels at screening: ≥ 1.40 and ≤ 5.60 mmol/L
* Fasting LDL-C levels at screening: ≥ 3.4 and ≤ 4.9 mmol/L

Exclusion Criteria:

* Recently (<6 months) diagnosed with cardiovascular event(s), revascularization or systemic inflammatory conditions.
* Medical history which might impact study measurements, to be judged by the study physician
* Use of over-the-counter and prescribed medication which may interfere with study measurements
* Reported weight loss or gain of 3 kg or more during a period of 2 months prior to screening.
* Currently smoking or being a non-smoker for less than 6 months and reported use of any nicotine containing products in the 6 months prior to screening and/or during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in TG concentrations | At baseline (after 2 weeks run-in period) and after 4 weeks intervention
  Two samples will be taken at baseline (Day -1 and 1) and two samples at the end of intervention (Day 28 and 29)

SECONDARY OUTCOMES:
Change in blood lipids | At baseline (after 2 weeks run-in period) and after 4 weeks intervention
  Two samples will be taken at baseline (Day -1 and 1) and two samples at the end of intervention (Day 28 and 29)

OTHER OUTCOMES:
Change in apolipoprotein concentrations | At baseline (after 2 weeks run-in period) and after 4 weeks intervention
  Samples will only be analyzed if relevant treatment effects on TG are observed

CONTACTS AND LOCATIONS:
Overall Officials: Wieneke Koppenol, MSc, Study Director — Unilever R&D
Locations (1):
- Charite Research Organisation, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blom WAM, Koppenol WP, Hiemstra H, Stojakovic T, Scharnagl H, Trautwein EA. A low-fat spread with added plant sterols and fish omega-3 fatty acids lowers serum triglyceride and LDL-cholesterol concentrations in individuals with modest hypercholesterolaemia and hypertriglyceridaemia. Eur J Nutr. 2019 Jun;58(4):1615-1624. doi: 10.1007/s00394-018-1706-1. Epub 2018 May 3. PMID 29725824